CLINICAL TRIAL: NCT06372990
Title: Development of a Rapid T-cell Analysis Test to Guide the Management of Patients With Chronic HBV and HBV/HDV Disease
Brief Title: Rapid T-cell Analysis Test in Patients With Chronic HBV and HBV/HDV Disease
Acronym: BDTc
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 0015338
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: HBV; HBV/HDV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBV: * 150 HBV patients under NUC treatment
  * 50 HBV patients with inactive carrier profile, treatment naive
- HBV/HDV: * 70 HDV patients treated with Bulevirtide
  * 30 HDV patients treatment naive

SUMMARY:
Prospective, non-pharmacological, single-center, non-profit observational study.

The study design allows longitudinal evaluation of the immune response during the natural history of the infection and/or treatment, correlating the data with the outcome of the disease and antiviral therapies, which will be collected as study variables from the source documents.

The study population will be patients suffering from chronic HBV infection with or without HBV-HDV co-infection followed at the Division of Gastroenterology and Hepatology of Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico.

The present study is part of an international cooperation project between the Division of Gastroenterology and Hepatology, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (Milan, Italy) and the Duke-NUS Medical School, Singapore, financed by a grant (project MAECI-2023-23683653) and divided into two specific Work Packages:

* WP 1 Milan team (WP1.1 - Clinical and virological phenotyping of CHB and CHD patients; WP1.2 - Clinical evaluation of rapid HBV T cell test in CHB and CHD populations)
* WP 2 Singapore team (WP2.1 - Applicability of the rapid T cell assay approach; WP 2.2 - Optimization of the rapid T cell assay protocol)

The primary objective of the study is to define the prevalence of specific T cell responses in patients with chronic HBV and HBV-HDV infection, through the application of a specific rapid T cell assay.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ability to understand and sign the informed consent
* chronic HBV infection or HBV-HDV co-infection defined by positivity of HBsAg antigen (HBV) and HDV RNA (HBV-HDV co-infection) for at least 6 months

Exclusion Criteria:

* Co-infection with other hepatotropic viruses (HCV, HIV)
* Treatment with immunosuppressive/immunomodulatory drugs
* Other congenital and/or acquired immunodeficiency conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol patients with chronic HBV infection (defined by HBsAg antigen positivity for at least 6 months) with or without HBV-HDV co-infection (defined by HDV RNA positivity for at least 6 months) who meet the inclusion criteria and do not present any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Define the prevalence of specific T cell responses in patients with chronic HBV and HBV-HDV infection, through the application of a specific rapid T cell assay | through study completion, an average of 2 year
  prevalence of HBV- and HDV-specific T cell responses in patients with chronic HBV infection with or without HBV-HDV co-infection

SECONDARY OUTCOMES:
Evaluate differences in terms of T cell response in patients with chronic HBV infection vs. HBV-HDV | through study completion, an average of 2 year
  differences in terms of T cell response in HBV vs. HBV-HDV
Correlate the T cell response phenotype with the clinical profile (chronic infection vs. chronic hepatitis), disease severity (cirrhosis vs. non-cirrhosis) and response to specific HBV and HBV-HDV therapies | through study completion, an average of 2 year
  correlation of the T cell response phenotype with the clinical profile (chronic infection vs. chronic hepatitis) and disease severity (cirrhosis vs. non-cirrhosis)
Improve the rapid T cell analysis protocol by simplifying the process, reducing analysis time and/or reducing the amount of material (blood) needed | through study completion, an average of 2 year
  development and optimization of a rapid method for performing immunological assays

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico, Division of Gastroenterology and Hepatology, Milan, Italy., Milan, MI, Italy